CLINICAL TRIAL: NCT04001946
Title: Clinical Trial of Gastrostomy Button Securement Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Collaborators: Phoenix Children's Hospital (Other); Stanford University (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-1615
Record Dates: First submitted 2019-05-08; First posted 2019-06-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-12

CONDITIONS: Gastrostomy Complications
Keywords: Gastrostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- G-button Securement Device (Other): Subjects will be provided instructions and a 12-week supply of test devices, sufficient to change the gauze dressing at least once per day.
  Interventions: Device: Button Huggie
- Standard Dressing (No Intervention): Subjects will be provided instructions and a 12-week supply of tape and gauze (current standard of care), sufficient to change the gauze dressing at least once per day.

INTERVENTIONS:
Device: Button Huggie — low profile, external securement device for G-buttons
  Arms: G-button Securement Device

SUMMARY:
Gastrostomy button (G-button) complications, such as granulation tissue formation, tube dislodgements, leakage, skin irritation or infection are frequent causes of post-operative clinic and emergency department visits. The investigators have developed a G-button securement device that they believe will have a significant reduction in the complications listed above. The investigators plan to randomized 200 patients to either the new securement device (treatment group) or the standard dressing (control group).

DETAILED DESCRIPTION:
Gastrostomy button (G-button) is a small tube inserted into the stomach that is used to feed and provide medication to children who can not eat or take medication on their own. G-buttons are commonly placed through surgery. While G-buttons give access for caregivers to provide adequate nutrition, they also can have complications associated with them; including, but not limited to leakage, skin irritation or infection, and dislodgement. These complications can be a big burden for caregivers and medical providers causing extra clinic, ED visits, and increased cost. The investigators have designed a securement device for the gastrostomy button and want to compare the device to the standard securement method, which is tape and gauze dressing. The investigators believe that they will show a significant reduction in the complications listed above. The investigators plan to randomized 200 patients to either the new securement device (treatment group) or the standard dressing (control group). The investigators plan to get feedback from caregivers at 4, 8, and 12 weeks. The G-button securement device that is a Class II, 510(k) exempt medical device, subject to General Controls under Product Code PLI, regulated by 21 CFR 876.5980.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 31 days to 18 years old who present for surgical placement of a gastrostomy button (open, endoscopically, or laparoscopically).
* Any patient with a pre-existing G-button who presents to the G-button or surgery clinic for G-button replacement or have complications associated with the G-button at any of study site locations.
* Patients admitted to the hospital with a pre-existing G-button for reasons unrelated to the G-button will be eligible for the study if they have complications with their current G-button site.

Exclusion Criteria:

* Refusal who object at any time to participate in the study
* Those whose parents or legal guardians cannot be reached by telephone
* Prisoners
* Pregnant women
* Impaired decision making capacity

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in G-button complications | entire study (3 months after placement)
  leakage, dislodgment, granulation tissue formation, and skin infection/irriation

SECONDARY OUTCOMES:
Caregiver Strain Index | entire study (3 months after placement)
  Obtain feedback from parents and patients at four, eight, and twelve weeks on various aspects of the securement device Comfort, quality of materials, adhesiveness, ease of use, types and number of interactions with healthcare providers (phone calls, ED, and clinic visits)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Phoenix Children's, Phoenix, Arizona
  - Stanford Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ezalife.com